CLINICAL TRIAL: NCT02712788
Title: Milrinone in Addition to Hyperdynamic Therapy in the Treatment of Vasospasm Following Aneurysmal Subarachnoid Hemorrhage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Completion not feasible due to lack of eligible subjects.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Scott Shapiro, MD, Professor of Neurological Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1505714749
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Vasospasm
Keywords: Subarachnoid Hemorrhage; Cerebral Vasospasm; Milrinone; Hyperdynamic Therapy
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage | interventions — Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milrinone (Active Comparator): Milrinone will be administered intravenously at an initial rate of 0.75mCg/kg/min and titrated based on symptoms in addition to hyperdynamic therapy and angiographic therapy as indicated per institutional protocol.
  Interventions: Drug: Milrinone
- Placebo (Placebo Comparator): Placebo (Normal Saline) will be administered intravenously and titrated based on symptoms in addition to hyperdynamic therapy and angiographic therapy as indicated per institutional protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milrinone
  Arms: Milrinone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the usefulness of adding Milrinone to the current standard treatment for cerebral vasospasm.

DETAILED DESCRIPTION:
The goal of this study is to assess the efficacy of milrinone as an agent to treat cerebral vasospasm by adding it to standard therapy. This will take the form of a randomized, controlled trial in which patients will receive either standard hyperdynamic therapy or hyperdynamic therapy + milrinone. The hypothesis of this study is that good outcomes will be 25% more common in the experimental (milrinone) group than the control (standard therapy) group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age
* Aneurysmal subarachnoid hemorrhage, proven on CT angiogram or digital subtraction angiography
* Aneurysm treated, either by endovascular embolization or surgical clip ligation
* Evidence of increased velocities on transcranial dopplers (TCDs) and/or radiographic evidence of vasospasm as seen on angiogram
* Cerebral vasospasm as demonstrated by patient's clinical exam (new focal deficit or change in mental status not attributable to any other cause)

Exclusion Criteria:

* Recurrent subarachnoid hemorrhage
* Untreated ruptured aneurysm, for any reason
* Patients who die prior to treatment for aneurysm
* Patients who are not able to complete at least 6 months of follow-up
* Patients who are admitted already in vasospasm (i.e. a delayed admission)
* Creatinine clearance less than 20 ml/min
* Women with a positive pregnancy test or who are lactating
* Other comorbidity which may adversely affect patient outcome, at the discretion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shapiro, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Heath Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abla AA, Wilson DA, Williamson RW, Nakaji P, McDougall CG, Zabramski JM, Albuquerque FC, Spetzler RF. The relationship between ruptured aneurysm location, subarachnoid hemorrhage clot thickness, and incidence of radiographic or symptomatic vasospasm in patients enrolled in a prospective randomized controlled trial. J Neurosurg. 2014 Feb;120(2):391-7. doi: 10.3171/2013.10.JNS13419. Epub 2013 Dec 6. PMID 24313610
- [Background] Diringer MN, Bleck TP, Claude Hemphill J 3rd, Menon D, Shutter L, Vespa P, Bruder N, Connolly ES Jr, Citerio G, Gress D, Hanggi D, Hoh BL, Lanzino G, Le Roux P, Rabinstein A, Schmutzhard E, Stocchetti N, Suarez JI, Treggiari M, Tseng MY, Vergouwen MD, Wolf S, Zipfel G; Neurocritical Care Society. Critical care management of patients following aneurysmal subarachnoid hemorrhage: recommendations from the Neurocritical Care Society's Multidisciplinary Consensus Conference. Neurocrit Care. 2011 Sep;15(2):211-40. doi: 10.1007/s12028-011-9605-9. PMID 21773873
- [Background] Fraticelli AT, Cholley BP, Losser MR, Saint Maurice JP, Payen D. Milrinone for the treatment of cerebral vasospasm after aneurysmal subarachnoid hemorrhage. Stroke. 2008 Mar;39(3):893-8. doi: 10.1161/STROKEAHA.107.492447. Epub 2008 Jan 31. PMID 18239182
- [Background] Lannes M, Teitelbaum J, del Pilar Cortes M, Cardoso M, Angle M. Milrinone and homeostasis to treat cerebral vasospasm associated with subarachnoid hemorrhage: the Montreal Neurological Hospital protocol. Neurocrit Care. 2012 Jun;16(3):354-62. doi: 10.1007/s12028-012-9701-5. PMID 22528278
- [Background] Nishiguchi M, Ono S, Iseda K, Manabe H, Hishikawa T, Date I. Effect of vasodilation by milrinone, a phosphodiesterase III inhibitor, on vasospastic arteries after a subarachnoid hemorrhage in vitro and in vivo: effectiveness of cisternal injection of milrinone. Neurosurgery. 2010 Jan;66(1):158-64; discussion 164. doi: 10.1227/01.NEU.0000363153.62579.FF. PMID 20023546

RESULTS

PARTICIPANT FLOW:
Groups:
- Milrinone: Milrinone will be administered intravenously at an initial rate of 0.75mCg/kg/min and titrated based on symptoms in addition to hyperdynamic therapy and angiographic therapy as indicated per institutional protocol.
  Milrinone
- Placebo: Placebo (Normal Saline) will be administered intravenously and titrated based on symptoms in addition to hyperdynamic therapy and angiographic therapy as indicated per institutional protocol.
  Placebo
Period: Overall Study
Arm/Group | Milrinone | Placebo
Started | 2 | 2
Completed | 0 | 2
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milrinone | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale (mRS) at 6 Months
Description: Reported as number for each subject and then will look statistically to see if there is a difference between the active arm and the placebo arm. The Modified Rankin scale is Scored as follows: 0 = No symptoms, 1 = No significant disability. Able to carry out all usual activities, despite some symptoms, 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability. Requires some help, but able to walk unassisted, 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent, 6 = Death. Higher scores indicate worse outcome.
Time Frame: 6 months
Population: The 2 subjects in the milrinone arm were unable to be analyzed. 1 subject was withdrawn due to ineligibilty and the other was withdrawn per physician discretion.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Milrinone | Placebo
Number analyzed (Participants) | 0 | 2
score on a scale |  | 1.5 [0 to 3]

2. Secondary Outcome: mRS at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Population: The 2 subjects in the milrinone arm were unable to be analyzed. 1 was withdrawn due to ineligibility and the other was withdrawn due to physician discretion.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Milrinone | Placebo
Number analyzed (Participants) | 0 | 2
score on a scale |  | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: 30 days following discontinuation of study drug
Arm/Group | Milrinone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milrinone (N=2) | Placebo (N=2)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Gastroduodenal Artery Bleed (Vascular disorders) | 1 (1) | 0 (0)
Thalamic and basal ganglia infarcts (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milrinone (N=2) | Placebo (N=2)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Fever (neurogenic) (Nervous system disorders) | 0 (0) | 1 (1)
epistaxis (Vascular disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute Deep Venous Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incontinence associated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02712788/Prot_SAP_000.pdf